CLINICAL TRIAL: NCT02402634
Title: Inflammatory Gene Polymorphism and Prolonged Mechanical Ventilation After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0989
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Patients With Postoperative Mechanical Ventilation After Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mechanical ventilatory lung care: liver transplantation recipients under mechanical ventilatory lung care
  Interventions: Other: Mechanical ventilatory lung care

INTERVENTIONS:
Other: Mechanical ventilatory lung care

SUMMARY:
Mechanical ventilatory lung care is essential for postoperative care in liver transplantation recipients, for such patients are under massive fluid challenge and hemodynamic alterations perioperatively. Some of the recipients experience difficulty in weaning off from the mechanical ventilator due to various causes. This study is to investigate the relationship between the inflammatory gene polymorphism, known for acute lung injury, and the duration of mechanical ventilatory care for such liver transplantation recipients.

ELIGIBILITY:
Inclusion Criteria:

1. 20-65 years old
2. scheduled for liver transplantation

Exclusion Criteria:

1. Patients under mechanical ventilation prior to surgery
2. patients with muscular skeletal disorder, probable cause for respiratory depression
3. patients not able to read, or understand the consent form
4. ethnicity, other than asian
5. patients refusal

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20-65 years old, scheduled for liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
total duration of postoperative ventilator care | an expected average of 2-3 days
  Time for successful weaning from ventilator could correlate with the inflammtory gene polymorphism, especially those related to acute lung injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea